CLINICAL TRIAL: NCT04575805
Title: Internet-delivered Combined Cognitive Bias Modification (iCBM-C) in People With High Obsessive Compulsive Symptoms: A Factorial Randomised Controlled Trial
Brief Title: Internet-delivered CBM-C for OC-symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sıla Derin, MA, Cilinical Psychologist, MA, Dokuz Eylul University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 120K044
Record Dates: First submitted 2020-09-26; First posted 2020-10-05 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Obsessive-compulsive Disorders and Symptoms; Obsessive Thoughts; Obsessive Compulsive Behavior
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Behavior

STUDY DESIGN:
Intervention Model Description: Factor 1: Cognitive Bias Modification-Interpretation (yes or no)
  Factor 2: Cognitive Bias Modification-Attention (yes or no)
  Each participant will be randomized to one of four conditions:
  Condition 1: Cognitive Bias Modification-Interpretation and Cognitive Bias Modification-Attention
  Condition 2: Cognitive Bias Modification-Interpretation and No Cognitive Bias Modification-Attention
  Condition 3: No Cognitive Bias Modification-Interpretation and Cognitive Bias Modification-Attention
  Condition 4: No Cognitive Bias Modification-Interpretation and No Attention Bias Modification-Attention
Who Masked: Participant
Masking Description: The participants will know that they will receive a treatment, but they will be blinded to randomization, i.e. will not know which groups they can be randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Internet-delivered Combined Cognitive Bias Modification (Experimental): CBM Version 1 is the combination of internet-delivered Cognitive Bias Modification-Interpretation and internet-delivered Cognitive Bias Modification-Attention interventions taking place over 4 weeks (eight sessions, twice per week).
  Interventions: Behavioral: Internet-delivered Combined Cognitive Bias Modification (iCBM-C)
- Internet-delivered Cognitive Bias Modification-Interpretation (Experimental): CBM Version 2 is an internet-delivered Cognitive Bias Modification-Interpretation intervention taking place over 4 weeks (eight sessions, twice per week).
  Interventions: Behavioral: Internet-delivered Cognitive Bias Modification-Interpretation (iCBM-I)
- Internet-delivered Cognitive Bias Modification-Attention (Experimental): CBM Version 3 is an internet-delivered Cognitive Bias Modification-Attention intervention taking place over 4 weeks (eight sessions, twice per week).
  Interventions: Behavioral: Internet-delivered Cognitive Bias Modification-Attention (iCBM-A)
- Wait-List Control (No Intervention): This arm is wait-list control group which will also receive internet-delivered Combined Cognitive Bias Modification intervention after the follow-up assessment

INTERVENTIONS:
Behavioral: Internet-delivered Combined Cognitive Bias Modification (iCBM-C) — The iCBM-C is online CBM intervention which is the combination of iCBM-I and iCBM-A interventions for obsessive-compulsive symptoms delivered in eight sessions, twice per week for 4 weeks. The presentation order of the two intervention components will be counterbalanced to allow exploration of any order effects. Thereby, half of the participants in iCBM-C group will complete the iCBM-A task followed by iCBM-I, while the other half will complete the iCBM-I task followed by iCBM-A during each session.
  Arms: Internet-delivered Combined Cognitive Bias Modification
Behavioral: Internet-delivered Cognitive Bias Modification-Interpretation (iCBM-I) — The iCBM-I is online CBM intervention for obsessive-compulsive symptoms comprised of delivery of OCD related scenarios taking place over eight sessions, twice per week for 4 weeks.
  Arms: Internet-delivered Cognitive Bias Modification-Interpretation
Behavioral: Internet-delivered Cognitive Bias Modification-Attention (iCBM-A) — The iCBM-A is online CBM intervention for obsessive-compulsive symptoms comprised of delivery of the modified dot-probe task taking place over eight sessions, twice per week for 4 weeks.
  Arms: Internet-delivered Cognitive Bias Modification-Attention

SUMMARY:
A factorial randomised controlled trial comparing internet-delivered combined cognitive bias modification intervention (iCBM-C) versus internet-delivered CBM-interpretation intervention (iCBM-I), internet-delivered CBM-attention intervention (iCBM-A) and wait-list control on obsessive-compulsive (OC) symptoms, OC-beliefs, OC-related interpretation and attention biases

DETAILED DESCRIPTION:
Cognitive behavioral therapy, consisting of exposure and response prevention and cognitive restructuring, is still one of the most effective treatments for obsessive compulsive disorder. However, some patients do not fully benefit from the treatment. This condition results in more search for novel approaches that can contribute to effectiveness of standard treatments. In this regard, the use of technology-based methods in recent researches is noteworthy. Cognitive bias modification (CBM) is one of these current efforts of technology-based methods. CBM involves computerized tasks designed to modify some cognitive biases such as attention and interpretation associated with psychopathology, particularly anxiety disorders. Researches have generally demonstrated that cognitive bias modification can be effective way to alter cognitive biases and to reduce anxiety symptoms. In recent years, there have been also some studies to investigate the potential effects of cognitive bias modification for obsessive compulsive disorder.The results of both CBM-Interpretation (CBM-I) and CBM-Attention (CBM-A) studies have shown that it is an effective and promising method in reducing cognitive biases in obsessive compulsive disorder (OCD). Although these studies are highly informative, they do not provide information about the causal role one bias has during the operation of another. In recent years, there has been a growing consensus that both biases arise from the same system, thereby, it is possible that modifying the system to alter one bias (e.g., attention), will also impact on the presence of the other bias.). In line with this notion, there are a couple of studies to test the effect of Combined Cognitive Bias Modification (CBM-C) which is combination of both CBM-A and CBM-I in intervention programs. The results of these studies are generally very positive. Although it is well established that attention bias and interpretation bias each have a key role in the development and maintenance of OCD, only one bias is targeted in CBM studies of OCD. Considering that a "combined cognitive bias" may contribute to the maintenance of several disorders, in order to try to maximise the potential clinical impact, the present research aims at exploring whether the combination of the CBM-A and CBM-I procedures would be more effective in reducing cognitive biases and OC symptoms than either alone. It is expected that internet-delivered CBM-C (iCBM-C) will result in superior treatment outcomes as indexed by internet-delivered CBM-I intervention only (iCBM-I), internet-delivered CBM-A intervention only (iCBM-A), and wait-list control (WLC).

ELIGIBILITY:
Inclusion Criteria:

* Fluent in written and spoken Turkish
* Daily access to the internet by computer
* No participation on any other interventional study or clinical trial
* The presence of high obsessive compulsive symptoms (Turkish version of Padua Inventory-Washington State University Revision scores > 65.81).

Exclusion Criteria:

* The absence of high obsessive compulsive symptoms (Turkish version of Padua Inventory-Washington State University Revision scores < 65.81)
* Suicidal ideation and severe psychotic symptoms (a rating of slight (i.e., 1) or greater on any item within the domain based on their responses to The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Self-Rated Level 1 Cross-Cutting Symptom Scale-Adult Version
* No access to the internet and computer
* Color blindness
* A current diagnosis of neurological and psychiatric disorder
* Ongoing psychological/psychiatric treatment
* Ongoing participation in other interventional study or clinical trial

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Padua Inventory-Washington State University Revision | Screen, Baseline (pre-intervention), post-intervention at week 4, 1-month follow-up
  Self-report questionnaire of obsessive compulsive symptoms composed of 39 items on a 5-point scale. Total score ranges from 0 to 156. Higher scores indicate greater severity of obsessive-compulsive symptoms (worse outcome).
Change in Obsessive Beliefs Questionnaire-44 | Baseline (pre-intervention), post-intervention at week 4, 1-month follow-up
  Self-report questionnaire of maladaptive obsessive-compulsive beliefs composed of 44 items on a 7-point scale. Total score ranges from 44 to 308. Higher score indicates that the individual has more maladaptive obsessive-compulsive beliefs (worse outcome).
Change in OC bias index | Baseline (pre-intervention), post-intervention at week 4
  Measure of interpretation biases. It is a computerized task that requires participants to read and imagine themselves in 10 OC-relevant test scenarios and 10 non OC-relevant scenarios with a title and missing letter in the final word of the sentence. Participants are then provided with a recognition rating form where they see the title of only the 10 OC-relevant scenarios in which they had previously imagined themselves. Each title corresponds with four different interpretations; target bias (OC-Positive and OC-Negative), and foil bias (Foil Positive and Foil Negative). Participants are asked to rate (on a 4-point scale) each sentence independently in terms of how similar each interpretation option is to the meaning of the scenario they had previously read. Target and Foil Bias Index scores are calculated by subtracting ratings for negative items from ratings for positive items. A positive score indicates that the individual has more OC-positive interpretations (better outcome).
Change in dot-probe task | Baseline (pre-intervention), post-intervention at week 4
  Measure of attention biases. Participants are presented 48 trials comprising all combinations of probe type ("←" or "→"), probe position (top or bottom), and picture type (neutral or threat). Each trial begins with the presentation of a central fixation cross for 500 ms. The cross is then replaced by a picture pair presented in the center of the screen for 500ms. After 500 ms, both stimuli disappear and a probe is shown in the location of one of the stimuli. Participants are instructed to indicate as quickly as possible which probe was shown via using keyboardResponse latencies are averaged to provide a single mean reaction time score for each participant. Scores are calculated by subtracting response latencies for trials in which the probe replaces threat stimuli from response latencies for trials in which the probe replaces neutral stimuli. subtracting the average. A negative bias score indicates an attention bias away from threat-related pictures (better outcome).

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scale-21 | Baseline (pre-intervention), post-intervention at week 4, 1-month follow-up
  Self-report questionnaire of the negative emotional states of depression, anxiety and stress composed of 21 questions on a 4-point scale. There are three subscales; (1) depression, (2) anxiety, and (3) stress. There are seven items in each of the subscales; the score of which ranges from 0 to 21. Higher scores indicate greater depression, anxiety anda stress (worse outcome).
Change in Positive and Negative Affect Schedule | Baseline (pre-intervention), post-intervention at week 4, 1-month follow-up
  Self-report questionnaire of positive and negative affect composed of 20 items with 10 positive and 10 negative affective descriptors on a 5-point scale. The positive and negative affect scales each have a potential range of 10-50. Higher scores on positive affect scale indicate higher positive affect (better outcome) whereas Higher scores on negative affect scale indicate higher negative affect (worse outcome).

OTHER OUTCOMES:
Feedback Form Questionnaire | post-intervention at week 4
  Measure of intervention acceptability and credibility. As well as items that are rated on continuous scales, there are open-ended questions to provide feedback on aspects they found helpful, unhelpful, liked, disliked and general improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Sıla Derin, MA, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No